CLINICAL TRIAL: NCT05917275
Title: Multi-Omics to Predict the Blood Pressure Response to Antihypertensives
Acronym: HT-PREDICT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 114516; 2023-505239-10-00 (Other: CTIS)
Record Dates: First submitted 2023-06-06; First posted 2023-06-23 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Amlodipine; olmesartan; Hydrochlorothiazide; Amlodipine Besylate, Olmesartan Medoxomil Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 4 weeks of Amlodipine (Experimental)
  Interventions: Drug: Amlodipine
- 4 weeks of Olmesartan (Experimental)
  Interventions: Drug: Olmesartan
- 4 weeks of Hydrochlorothiazide (Experimental)
  Interventions: Drug: Hydrochlorothiazide
- 4 weeks of Amlodipine/Olmesartan (Experimental)
  Interventions: Drug: Amlodipine/Olmesartan

INTERVENTIONS:
Drug: Amlodipine — 4 weeks of Amlodipine
  Arms: 4 weeks of Amlodipine
Drug: Olmesartan — 4 weeks of Olmesartan
  Arms: 4 weeks of Olmesartan
Drug: Hydrochlorothiazide — 4 weeks of Hydrochlorothiazide
  Arms: 4 weeks of Hydrochlorothiazide
Drug: Amlodipine/Olmesartan — 4 weeks of Amlodipine/Olmesartan
  Arms: 4 weeks of Amlodipine/Olmesartan

SUMMARY:
The goal of this clinical trial is to develop biomarkers composed of multiple OMICs (MOMICs) for prediction of blood pressure response to antihypertensive drugs in the treatment of primary hypertension. The main objectives are:

* Primary objective:

  - To identify MOMICs biomarkers that predict the response in 24-hour blood pressure to antihypertensive treatment for each treatment group (olmesartan, amlodipine, hydrochlorothiazide, olmesartan/amlodipine)
* Secondary objectives:

  * To identify a MOMICs biomarker that predict the response in night-time blood pressure to anti-hypertensive treatment for each treatment group (olmesartan, amlodipine, hydrochlorothiazide, olmesartan/amlodipine)
  * To identify MOMICs biomarkers that predict side effects, including changes in QoLof olmesartan, amlodipine and hydrochlorothiazide.
* Exploratory objective:

  * To assess changes in MOMICs biomarkers induced by each drug

Participants will undergo three 4-week treatment periods:

* Each subject receives 3 out of 4 possible treatments (olmesartan, amlodipine, hydrochlorothiazide, olmesartan/amlodipine).
* Before and after each treatment period OMICS measurements and an ABPM are performed.
* At the end of each treatment period blood is sampled for drug level testing to assess adherence.
* Electrolytes and kidney function are checked 5-7 days after start of each treatment period.

ELIGIBILITY:
Inclusion criteria

* Age 18 up to and including 75 years
* 24 hours systolic blood pressure 130-164 (corresponding with grade 1-2 hypertension), without the use of blood pressure lowering agents (at screening for patients without pre-treatment or after 4 week wash-out of antihypertensive medication for subjects using a single antihypertensive agent at screening)
* Indication for antihypertensive therapy according to the 2023 European Society of Hypertension Guidelines for the management of arterial hypertension
* Subject is not treated with antihypertensive drugs or is treated with a single antihypertensive drug.
* Female patients must be non-lactating and at no risk of pregnancy for one of the following reasons: 1 year postmenopausal, surgically sterile, or willing to use an acceptable method of contraception (oral contraceptives, approved contraceptive implants, long-term injectable contraception, intrauterine devices, or tubal ligation are allowed.)

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Treatment with 2 or more antihypertensive drugs < 3 months before inclusion. It is not allowed to stop medication for study purposes in subjects treated with 2 or more anti-hypertensive drugs.
* Known diagnosis of secondary hypertension to an identifiable cause other than treated sleep apnea (e.g., hyperaldosteronism, renal artery stenosis, pheochromocytoma, Cushing's syndrome, coarctation of the aorta, uncontrolled hyper- or hypothyroidism and intracranial tumor)
* Use of VEGF inhibitors, calcineurin inhibitors, glucocorticosteroids, erythropoietin stimulation agents, daily use of NSAID's
* Use of MDMA, methamphetamine, cocaine
* Use of glycyrrhetinic acid containing products , i.e. liquorice, specific herbal teas, <4 weeks before inclusion. (If patients are willing to stop the intake of glycyrrhetinic acid containing products for the duration of the trial, they can be rescreened after 4 weeks of stopping glycyrrhetinic acid containing products)
* Use of potassium containing supplements
* Concurrent use of medication or a supplement with significant drug interaction with study medication. Special attention is warranted for amlodipine which is metabolized by Cyp3A4. Subjects using strong inhibitors or inducers of Cyp3A4 are excluded from participation in this trial. A list of strong inhibitors and inducers is provided in Addendum 1 of this protocol. For information on possible drug interactions we refer to the website of Lexi-Interact Online (Lexicomp® Drug Interactions - UpToDate (doctorabad.com): https://doctorabad.com/UpToDate/d/di.htm).
* History of myocardial infarction, angina pectoris
* History of atrial fibrillation
* History of severe valvular or structural heart disease (excluding left ventricular hypertrophy)
* History of NYHA class III or IV heart failure or known reduced left ventricular function (ejection fraction (EF) <30%)
* History of cerebrovascular accident or transient ischemic attack
* History of hypertensive crisis
* History of liver failure
* History of skin cancer
* History of gout
* Current hyperparathyroidism
* Current biliary tract obstruction
* Pregnancy
* Life expectancy < 1 year
* Known side effect or contra-indication to treatment with calcium channel blockers
* Known side effect or contra-indication to treatment with angiotensin II receptor blockers
* Known side effect or contra-indication to treatment with thiazide diuretics
* Arm circumference > 46 cm
* Sodium level outside reference range at screening visit
* Potassium level outside reference range at screening visit
* Calcium level outside reference range at screening visit
* eGFR < 50 ml/min/1,73m2
* Use of loop diuretics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Predictive value of Multi-Omics profile for blood pressure | 4 weeks after start treatment
  Predictive value of a MOMICs profile to discriminate subjects with a decrease in 24-hour blood pressure below the median from subjects with a decrease in 24-hour blood pressure above the median for each treatment group (olmesartan, amlodipine, hydrochlorothiazide, olmesartan/amlodipine).

SECONDARY OUTCOMES:
Predictive value of Multi-Omics profile for night-time blood pressure | 4 weeks after start treatment
  Predictive value of a MOMICs profile to discriminate subjects with a decrease in night-time blood pressure below the median from subjects with a decrease in 24-hour blood pressure above the median, for each treatment group (olmesartan, amlodipine, hydrochlorothiazide, olmesartan/amlodipine).
Correlation Multi-Omics profile and adverse effects | correlation between changes from baseline to 4 weeks after start treatment
  Correlation between changes in individual biomarkers and adverse effects as documented using adverse effects questionnaire and SF-36

OTHER OUTCOMES:
Changes in Multi-Omics profile after treatment | 4 weeks after start treatment
  Change in individual Multi-Omics profile components after treatment with olmesartan, amlodipine and hydrochlorothiazide compared with biomarkers levels at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Joost Rutten, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No